CLINICAL TRIAL: NCT02858908
Title: A Single-Blind, Phase 2 Study To Evaluate The Safety And Efficacy Of Tideglusib 400mg Or 1000mg For The Treatment Of Adolescent And Adult Congenital And Juvenile-Onset Myotonic Dystrophy
Brief Title: Study of Tideglusib in Adolescent and Adult Patients With Myotonic Dystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AMO Pharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: AMO-02-MD-2-001; 2016-000067-16 (EudraCT Number)
Expanded Access: NCT07119775 (Available)
Record Dates: First submitted 2016-08-04; First posted 2016-08-08 (Estimated); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Myotonic Dystrophy 1
MeSH Terms: conditions — Myotonic Dystrophy | interventions — tideglusib

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 - Tideglusib (Experimental): 1000 mg tideglusib, orally, once daily
  Interventions: Drug: Tideglusib
- Cohort 2 - Tideglusib (Experimental): 400 mg tideglusib, orally, once daily
  Interventions: Drug: Tideglusib

INTERVENTIONS:
Drug: Tideglusib — Tideglusib for oral suspension,

SUMMARY:
The purpose of this study is to determine whether Tideglusib is safe and efficacious in the treatment of adolescents and adults with congenital and juvenile-onset Myotonic Dystrophy. The pharmacokinetics of tideglusib and its primary metabolite will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents or adults with diagnosis of congenital or juvenile-onset type 1 myotonic dystrophy (DM-1)
* Diagnosis must be genetically confirmed
* Subjects must be male or female aged 12 years to 45 years
* Subjects must have a Clinical Global Impression - Severity (CGI-S) score of 4 or greater at Screening and Run-in (V2)
* Subjects must be ambulatory and able to complete the 10 metre walk/run test (splints allowed)
* Subject's legally authorized representative (LAR) must provide written informed consent and there must be written consent or assent (as age applicable and developmentally appropriate) by the subject before any study-related procedures are conducted

Exclusion Criteria:

* Non-ambulatory (full time) wheel chair user
* Receiving stimulant medication
* Receiving other medications/therapies not stable (changed) within 4 weeks prior to Run-in (V2)
* Medical illness or other concern which would cause investigator to conclude subjects will not be able to perform the study procedures or assessments or would confound interpretation of data obtained during assessment.
* Current enrolment in a clinical trial of an investigational drug or enrolment in a clinical trial of an investigational drug in the last 6 months
* Women of child bearing potential who are pregnant, lactating or not willing to use a protocol defined acceptable contraception method if sexually active and not surgically sterile.
* Gastrointestinal disease which may interfere with the absorption, distribution, metabolism or excretion of the study medication and impact the interpretability of the study results
* Current clinically significant (as determined by the investigator) cardiovascular, renal, hepatic, endocrine or respiratory disease
* Clinically significant heart disease (in the opinion of the investigator) or second or third degree heart block, atrial flutter, atrial fibrillation, ventricular arrhythmias, or is receiving medication for treatment of a cardiac arrhythmia
* A history of chronic liver disease with current out of range values for Alanine transaminase (ALT), clinically relevant hepatic steatosis or other clinical manifestations of ongoing liver disease
* A history of significant drug allergy (such as Steven-Johnson syndrome, anaphylaxis)
* A history of alcohol or substance use disorders

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grainne Gorman, MB BCh BAO LRCP&SI MRCP FRCP, Principal Investigator — Institute of Neuroscience, Newcastle University.
Locations (1):
- Newcastle-upon-Tyne Hospitals NHS Trust, Newcastle upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- [Derived] Horrigan J, Gomes TB, Snape M, Nikolenko N, McMorn A, Evans S, Yaroshinsky A, Della Pasqua O, Oosterholt S, Lochmuller H. A Phase 2 Study of AMO-02 (Tideglusib) in Congenital and Childhood-Onset Myotonic Dystrophy Type 1 (DM1). Pediatr Neurol. 2020 Nov;112:84-93. doi: 10.1016/j.pediatrneurol.2020.08.001. Epub 2020 Aug 5. PMID 32942085

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were to be male or female aged 12 to 45 years with a diagnosis of genetically confirmed congenital or juvenile-onset type 1 myotonic dystrophy. Subjects were to have a Clinical Global Impression- Severity (CGI-S) score of 4 or greater at Screening and Run-in (V2) and were to be ambulatory and able to complete the 10-metre walk/run test.
Groups:
- Cohort 1: Subjects were given tideglusib 1000 mg for 12 weeks (weeks 0 to 12)
- Cohort 2: Subjects were given tideglusib 400 mg for 12 weeks (weeks 0 to 12)
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: 1000 mg tideglusib
- Cohort 2: 400 mg tideglusib
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Customized [Mean (Standard Deviation); unit: years]
  Mean | 21.8 (5.5) | 20.3 (6.36) | 21 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 3 | 7 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or latino | 8 | 8 | 16
  White | 8 | 7 | 15
  Asian | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety (Adverse Events)
Description: Incidence of Adverse events (AEs), including serious adverse events (SAEs), between baseline to end of study.
Time Frame: 12 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Participants
  Total number of TEAEs | 8 | 6
  Total number of serious TEAEs | 0 | 0
  Total number of TEAEs leading to discontinuation of active treatment | 0 | 0
  Total number of TEAEs leading to withdrawal | 0 | 0
  Total number of TEAEs leading to death | 0 | 0
  Severity: Mild | 3 | 1
  Severity: Moderate | 5 | 4
  Severity: Severe | 0 | 1
  Unrelated to active treatment | 6 | 6
  Related to active treatment | 2 | 0

2. Secondary Outcome: Plasma Concentration of Tideglusib
Description: Pharmacokinetic samples were collected to determine Tideglusib plasma concentration
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
ng/mL
  Maximum plasma concentration (Cmax) | 1041.25 (361.44) | 496.94 (104.88)
  Minimum plasma concentration (Cmin) | 8.63 (5.68) | 5.14 (4.06)
  Steady-state concentration (CSS) | 133.7 (60.79) | 54.27 (16.54)

3. Secondary Outcome: Blood Pharmacokinetics of Tideglusib
Description: Pharmacokinetic samples were collected to determine time of the maximum plasma concentration and terminal elimination half-life of tideglusib
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
h
  Time of the maximum plasma concentration (Tmax) | 0.79 (0.27) | 0.65 (0.29)
  Terminal elimination half-life (T1/2) | 1.82 (0.64) | 2.68 (1.70)

4. Secondary Outcome: Area Under the Plasma Concentration vs. Time Curve of Tideglusib
Description: Pharmacokinetic samples were collected to determine area under the plasma concentration vs. time curve from 0 to 12 h and area under the plasma concentration vs. time curve from 0 to 24 h of tideglusib
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL.h
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
ng/mL.h
  Area under the plasma concentration vs. time curve from 0 to 12 h (AUC0-12) | 3054.27 (1418.30) | 1214.88 (390.81)
  Area under the plasma concentration vs. time curve from 0 to 24 h (AUC0-24) | 3208.8 (1459.03) | 1302.42 (396.96)

5. Secondary Outcome: 10 Metre Walk/Run Test
Description: The 10-metre walk/run test is a performance measure used to assess walking speed in metres per second over a short distance and was used as an assessment of functional mobility. Time taken to complete the 10m walk/run test at fastest and preferred speed is measured.
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
seconds
  Preferred speed (observed value at week 12) | 9.1041 (1.34351) | 9.1475 (1.72651)
  Preferred speed (change from baseline at week 12) | -0.6616 (1.96370) | -0.6529 (0.86109)
  Fastest speed (observed value at week 12) | 4.2515 (2.41439) | 4.4833 (2.72809)
  Fastest speed (change from baseline at week 12) | -0.3894 (0.32806) | -0.0650 (0.46428)
Statistical Analysis 1: Comparison: Cohort 1; Change from baseline to week 12 in the time taken (seconds) to complete 10-metre walk/run test at the preferred speed; Test type: Other — Analysis of change in efficacy variables from baseline to week 12 were performed using mixed effect model repeated measures (MMRM) with baseline value as a covariate, dose group and visit as fixed effects and a treatment-by-visit interaction. Adjusted least square mean estimates were produced by dose group and study visit and were presented with two-sided 95% confidence intervals and p-values; p = 0.0484, Mixed Models Analysis; Mean Difference (Net) = -0.6696, 95% CI 2-sided [-1.3340 to -0.0051] — The mean difference is an adjusted Least Square Mean
Statistical Analysis 2: Comparison: Cohort 2; Change from baseline to week 12 in the time taken (seconds) to complete 10-metre walk/run test at the preferred speed; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.0565, Mixed Models Analysis; Mean Difference (Net) = -0.6449, 95% CI 2-sided [-1.3094 to 0.0195] — The mean difference is an adjusted Least Square Mean

6. Secondary Outcome: Computerised Handgrip Myometer Measure of Grip Strength and Muscle Relaxation Time
Description: Handgrip myometry is used as a measure of myotonia and muscle strength for the dominant hand
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
kg
  Observed value (at week 12) | 14.0899 (7.71583) | 14.1334 (6.86499)
  Change from baseline (at week 12) | 1.0098 (3.09422) | -1.4893 (2.89328)
Statistical Analysis 1: Comparison: Cohort 1; Change from baseline to week 12 in grip strength (kg); Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.3732, Mixed Models Analysis; Mean Difference (Net) = 0.9102, 95% CI 2-sided [-1.1526 to 2.9730] — The mean difference is an adjusted Least Square Mean
Statistical Analysis 2: Comparison: Cohort 2; Change from baseline to week 12 in grip strength (kg); Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.1782, Mixed Models Analysis; Mean Difference (Net) = -1.3897, 95% CI 2-sided [-3.4525 to 0.6731] — The mean difference is an adjusted Least Square Mean

7. Secondary Outcome: Respiratory Forced Vital Capacity (FVC)
Description: FVC is a measure of lung function (the total amount of air exhaled during a Forced Expiratory Volume is measured using a spirometer)
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
litres
  Observed value (at week 12) | 2.1509 (0.93362) | 2.4220 (1.15969)
  Change from baseline (at week 12) | -0.0179 (0.32603) | 0.0118 (0.36746)
Statistical Analysis 1: Comparison: Cohort 1; Change from baseline to week 12 in FVC (litres); Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.8886, Mixed Models Analysis; Mean Difference (Net) = -0.0213, 95% CI 2-sided [-0.3368 to 0.2941] — The mean difference is an adjusted Least Square Mean
Statistical Analysis 2: Comparison: Cohort 2; Change from baseline to week 12 in FVC (litres); Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.9204, Mixed Models Analysis; Mean Difference (Net) = 0.0152, 95% CI 2-sided [-0.3003 to 0.3307] — The mean difference is an adjusted Least Square Mean

8. Secondary Outcome: Dual-energy X-ray Absorptiometry (DXA)
Description: DXA utilises two low energy X-ray beams, with different energy levels, which are aimed at the subject's bones. The DXA scan is more typically used to measure bone mineral density, however it can also be used to measure total lean muscle mass
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
gram
  Arms (observed value at week 12) | 3102.9 (898.69) | 4098.5 (1313.53)
  Arms (change from baseline at week 12) | -252.8 (1038.49) | 35.9 (357.09)
  Legs (observed value at week 12) | 11767.0 (2980.78) | 12262.8 (3225.63)
  Legs (change from baseline at week 12) | -62.5 (646.22) | 95.0 (299.82)
  Total (observed value at week 12) | 38267.6 (8274.58) | 37740.4 (8481.27)
  Total (change from baseline at week 12) | 411.6 (2040.84) | 391.9 (763.01)
Statistical Analysis 1: Comparison: Cohort 1; Changes from baseline to week 12 in the DXA scan total lean muscle mass (g); Test type: Other — The exact Wilcoxon signed rank test was used to test for a change in the DXA scan total lean muscle mass (g) from baseline to end of treatment; p = 1.0000, ANCOVA; Median Difference (Net) = -42.75, 95% CI 2-sided [-1270.00 to 2178.50] — Hodges-Lehmann estimates for the median and confidence intervals are presented
Statistical Analysis 2: Comparison: Cohort 2; Changes from baseline to week 12 in the DXA scan total lean muscle mass (g); Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.3125, ANCOVA; Median Difference (Net) = 426.75, 95% CI 2-sided [-289.50 to 1198.50] — Hodges-Lehmann estimates for the median and confidence intervals are presented

9. Secondary Outcome: Clinical Global Impressions- Severity (CGI-S)
Description: The CGI-S is a 7-point Likert type scale that requires the clinician to rate the severity of the subject's illness at the time of assessment, relative to the clinician's past experience with subjects who have the same diagnosis. Considering total clinical experience, a subject is assessed on severity of illness at the time of rating 1, normal, not at all ill; 2, borderline ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill. Change in CGI-S was observed in only 1 subject. Consequently statistical analysis was not conducted.
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Values on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Values on a scale
  Observed value at week 12 | 4.8 (1.16) | 4.9 (0.83)
  Change from baseline at week 12 | -0.1 (0.35) | 0.0 (0.00)

10. Secondary Outcome: Clinical Global Impressions- Improvement (CGI-I)
Description: The CGI-I requires the clinician to rate how much the subject's illness has improved or worsened relative to a baseline state.
  A seven point Likert type scale is used from 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, 7 = very much worse.
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Scores on a scale | 3.1 (0.83) | 3.0 (1.07)
Statistical Analysis 1: Comparison: Cohort 1; Observed value at week 12 in Clinical Global Impression Global Improvement Scale (CGI-I); Test type: Other — A mixed effect model repeated measure (MMRM) was fitted to the observed values at week12. The model included dose group and visit as fixed effects, and the treatment-by-visit interaction. F-tests from PROC MIXED were based on Kenward-Roger's adjusted degrees of freedom; p = 0.0030, Mixed Models Analysis — The p-value is presented for the comparison of adjusted Least Square Means to a score of 4, representing 'No change'; Mean Difference (Net) = 3.1, 95% CI 2-sided [2.6 to 3.7]
Statistical Analysis 2: Comparison: Cohort 2; Observed value at week 12 in Clinical Global Impression Global Improvement Scale (CGI-I); Test type: Other — [test comment as in outcome 10, analysis 1]; p = 0.0009, Mixed Models Analysis — The p-value is presented for the comparison of adjusted Least Square Means to a score of 4, representing 'No change'; Mean Difference (Net) = 3.0, 95% CI 2-sided [2.4 to 3.6]

11. Secondary Outcome: Actigraphy (3-minute Bouts of Activity)
Description: Actigraphy is a non-invasive method of monitoring physical activity via an actigraph device. The actigraph device was worn on the waist during waking hours, according to the device's instruction manual.
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: 3 minute bouts of activity per hour
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
3 minute bouts of activity per hour
  Weekly total number of 3 minute bouts of activity (observed value at week 12) | 1.465 (0.1780) | 0.938 (0.5268)
  Weekly total number of 3 minute bouts of activity (change from baseline at week 12) | -0.200 (0.3959) | -0.284 (0.1805)
Statistical Analysis 1: Comparison: Cohort 1; Change from baseline to week 12 in the weekly total number of 3 minute bouts of activity per hour wear time; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.1857, Mixed Models Analysis; Mean Difference (Net) = -0.132, 95% CI 2-sided [-0.330 to 0.066] — The mean difference is an adjusted Least Square Mean
Statistical Analysis 2: Comparison: Cohort 2; Change from baseline to week 12 in the weekly total number of 3 minute bouts of activity per hour wear time; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.0054, Mixed Models Analysis; Mean Difference (Net) = -0.325, 95% CI 2-sided [-0.549 to -0.102] — The mean difference is an adjusted Least Square Mean

12. Secondary Outcome: Actigraphy (>10-minute Bouts of Activity)
Description: as for outcome 11
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: 10 minute bouts of activity per hour
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
10 minute bouts of activity per hour
  Weekly total number of >10 minute bouts of activity (observed value at week 12) | 0.048 (0.0621) | 0.020 (0.0245)
  Weekly total number of >10 minute bouts of activity (change from baseline at week 12) | -0.010 (0.0600) | 0.006 (0.0313)

13. Secondary Outcome: Actigraphy (Steps)
Description: as for outcome 11
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: steps per hour wear time
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
steps per hour wear time
  Weekly total number of steps (observed value at week 12) | 556.387 (255.6433) | 352.518 (263.1992)
  Weekly total number of steps (change from baseline at week 12) | -51.427 (198.9754) | -53.802 (89.0843)

14. Secondary Outcome: Nine Hole Peg Test (NHPT)
Description: Measure of fine manual dexterity. Time to taken to complete the NHPT (dominant hand) is recorded.
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
seconds
  Observed value at week 12 | 23.590 (8.2592) | 24.760 (3.8275)
  Change from baseline at week 12 | -2.168 (3.9007) | -0.950 (1.7080)
Statistical Analysis 1: Comparison: Cohort 1; Change from baseline to week 12 in the time taken (seconds) to complete the nine hole peg test for the dominant arm; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.0111, Mixed Models Analysis; Mean Difference (Net) = -2.162, 95% CI 2-sided [-3.731 to -0.593] — The mean difference is an adjusted Least Square Mean
Statistical Analysis 2: Comparison: Cohort 2; Change from baseline to week 12 in the time taken (seconds) to complete the nine hole peg test for the dominant arm; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.2088, Mixed Models Analysis; Mean Difference (Net) = -0.955, 95% CI 2-sided [-2.525 to 0.614] — The mean difference is an adjusted Least Square Mean

15. Secondary Outcome: Top 3 Concerns Visual Analogue Scale (VAS) Score
Description: The Top 3 concerns VAS allows caregivers to identify their main three causes of concern, related to the subject's myotonic dystrophy, rather than these being pre-specified within a scale and then rating how these concerns have changed at specific time-points during the study. Subjects, where possible, and caregivers were asked to rate three causes for concern by drawing a vertical mark on a 10 cm long visual analogue scale with anchors of "not at all severe" at the left end (0 cm) and "very severe" at the right end (10 cm). A score for each concern was to be determined by measuring the number of centimeters on the 10 cm VAS line from the anchor point on the left side of the line. A total VAS score for each subject was calculated as the sum of the scores for the 3 concerns (minimum = 0 cm, maximum = 30 cm). A higher score represents a worse outcome.
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Score on a scale
  Subject Top 3 Concerns VAS total score (observed value at week 12) | 15.66 (6.331) | 15.29 (5.641)
  Subject Top 3 Concerns VAS total score (change from baseline at week 12) | -1.76 (3.455) | -2.00 (2.598)
  Caregiver Top 3 Concerns VAS total score (observed value at week 12) | 18.84 (3.583) | 16.58 (6.151)
  Caregiver Top 3 Concerns VAS total score (change from baseline at week 12) | -2.39 (2.669) | -1.98 (2.001)
Statistical Analysis 1: Comparison: Cohort 1; Change from baseline to week 12 in the subject top three concerns VAS total score (cm); Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.0728, Mixed Models Analysis; Mean Difference (Net) = -1.77, 95% CI 2-sided [-3.71 to 0.18] — The mean difference is an adjusted Least Square Mean
Statistical Analysis 2: Comparison: Cohort 2; Change from baseline to week 12 in the subject top three concerns VAS total score (cm); Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.0456, Mixed Models Analysis; Mean Difference (Net) = -1.99, 95% CI 2-sided [-3.94 to -0.04] — The mean difference is an adjusted Least Square Mean
Statistical Analysis 3: Comparison: Cohort 1; Change from baseline to week 12 in the caregiver top three concerns VAS total score (cm); Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.0058, Mixed Models Analysis; Mean Difference (Net) = -2.41, 95% CI 2-sided [-4.03 to -0.80] — The mean difference is an adjusted Least Square Mean
Statistical Analysis 4: Comparison: Cohort 2; Change from baseline to week 12 in the caregiver top three concerns VAS total score (cm); Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.0208, Mixed Models Analysis; Mean Difference (Net) = -1.95, 95% CI 2-sided [-3.56 to -0.34] — The mean difference is an adjusted Least Square Mean

16. Secondary Outcome: Ohio State University (OSU) Autism Rating Scale (OARS)
Description: The OARS-4 contains the autism signs and symptoms in the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition. These were to be rated with the degree of impairment the subject experiences for the given symptom. The symptoms were to be elicited in a semi-structured interview with the subject's primary caregiver. The assessor was to take both frequency/duration and degree of impairment into account and how much the item interferes with relationships, learning, and/or activities of daily living. The scores for this assessment were from 0 (Never or Rarely; Not a Problem) to 3 (Very Often; A Severe Problem): a score for each symptom of social impairment, communication impairment and restricted patterns were averaged to provide a total impairment score. A higher score represents a worse outcome (minimum = 0, maximum 3).
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Units on a scale
  Total impairment mean (observed value at week 12) | 0.239 (0.3178) | 0.303 (0.4946)
  Total impairment mean (change from baseline at week 12) | -0.054 (0.0782) | -0.010 (0.0283)
Statistical Analysis 1: Comparison: Cohort 1; Change from baseline to week 12 in the OSU Autism Rating Scale - DSM-IV (OARS-4) total impairment mean; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.0068, Mixed Models Analysis; Mean Difference (Net) = -0.054, 95% CI 2-sided [-0.092 to -0.017] — The mean difference is an adjusted Least Square Mean
Statistical Analysis 2: Comparison: Cohort 2; Change from baseline to week 12 in the OSU Autism Rating Scale - DSM-IV (OARS-4) total impairment mean; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.6090, Mixed Models Analysis; Mean Difference (Net) = -0.009, 95% CI 2-sided [-0.047 to 0.028] — The mean difference is an adjusted Least Square Mean

17. Secondary Outcome: Ohio State University (OSU) Autism Clinical Global Impression (CGI)
Description: The OSU Autism CGI scale contains separate subscales for symptom severity and for global improvement. These are rated in a similar way to the National Institute of Mental Health (NIMH) CGI Severity scale, but it is focused on autism spectrum symptoms. OSU Autism CGI-severity and OSU Autism CGI-improvement scores use a seven point Likert rating scale from 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, 7 = very much worse.
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Units on a scale
  OSU autism CGI-Severity (observed value at week 12) | 1.9 (0.99) | 2.3 (1.83)
  OSU autism CGI-Severity (change from baseline at week 12) | -0.1 (0.35) | 0 (0)
  OSU autism CGI-Improvement (observed value at week 12) | 3.4 (0.74) | 4 (0)
Statistical Analysis 1: Comparison: Cohort 1; Observed value at week 12 in OSU global improvement scale for autism (OSU CGI-I); Test type: Other — A mixed effect model repeated measure (MMRM) was fitted to the observed values at week12 in OSU CGI-I. The model included dose group and visit as fixed effects, and the treatment-by-visit interaction. F-tests from PROC MIXED were based on Kenward-Roger's adjusted degrees of freedom. A compound symmetry covariance matrix was used for the repeated visits within subject; p = 0.0011, Mixed Models Analysis — p-values are presented for the comparison of adjusted Least Square Means to a score of 4, representing 'No change'; Mean Difference (Net) = 3.4, 95% CI 2-sided [3.0 to 3.7]
Statistical Analysis 2: Comparison: Cohort 2; Observed value at week 12 in OSU global improvement scale for autism (OSU CGI-I); Test type: Other — [test comment as in outcome 17, analysis 1]; p = 1.0000, Mixed Models Analysis — p-values are presented for the comparison of adjusted Least Square Means to a score of 4, representing 'No change'; Mean Difference (Net) = 4.0, 95% CI 2-sided [3.6 to 4.4]

18. Secondary Outcome: Clinician-completed Domain Specific Cause for Concern Visual Analogue Scale (VAS): Myotonic Dystrophy
Description: The Clinician-completed Domain Specific Causes for Concern is a Visual Analogue Scale completed by the clinician that scores the severity of concerns of domains that are clinically relevant in myotonic dystrophy. The severity of the clinician's concern is scored by using a 10 cm visual analogue scale (VAS), with anchors of "not at all severe" at the left end (0 cm) and "very severe" at the right end (10 cm). The clinician is asked to make a vertical line indicating his/her level of concern in each domain, using a time frame of the past week for reference. A score is to be determined by measuring the number of centimeters on the 10 cm VAS line from the anchor point on the left side of the line. A total VAS score for each subject was calculated as the sum of the scores for the 17 domains (minimum = 0, maximum = 170 cm). A higher score represents a worse outcome.
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Score on a scale
  VAS total score (observed value at week 12) | 51.19 (8.798) | 59.28 (17.450)
  VAS total score (change from baseline at week 12) | -5.80 (4.855) | -3.38 (2.726)
Statistical Analysis 1: Comparison: Cohort 1; Change from baseline at week 12 in the clinician-completed domain specific causes for concern VAS total score (cm); Test type: Other — [test comment as in outcome 5, analysis 1]; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -5.91, 95% CI 2-sided [-8.35 to -3.47] — The mean difference is an adjusted Least Square Mean
Statistical Analysis 2: Comparison: Cohort 2; Change from baseline at week 12 in the clinician-completed domain specific causes for concern VAS total score (cm); Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.0116, Mixed Models Analysis; Mean Difference (Net) = -3.27, 95% CI 2-sided [-5.71 to -0.83] — The mean difference is an adjusted Least Square Mean

19. Secondary Outcome: Peabody Picture Vocabulary Test (PPVT)
Description: The PPVT-4 scale is a norm-referenced instrument for measuring the receptive (hearing) vocabulary of children and adults. It contains training items and 228 test items, each consisting of four full-colour pictures as response options on a page. For each item, the examiner says a word, and the examinee responds by selecting the picture that best illustrates that word's meaning. Each administration of the test produces a raw score (number of test items answered correctly), which can be converted to a standard score (using age-based norms) with a mean of 100 and a standard deviation of 15. Higher scores mean a better performance/receptive vocabulary.
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
Units on a scale
  Age-based standard score (observed value at week 12) | 63.8 (15.81) | 79.8 (22.23)
  Age-based standard score (change from baseline at week 12) | -0.1 (7.97) | -1.1 (5.57)
Statistical Analysis 1: Comparison: Cohort 1; Change from baseline to week 12 in the peabody picture vocabulary test age-based standard score; Test type: Other — An ANCOVA was fitted to the change in the Peabody Picture Vocabulary Test age-based standard score from baseline to end of treatment. The model included the baseline value as a covariate and dose group as a fixed effect; p = 0.6631, ANCOVA; Mean Difference (Net) = -1.1, 95% CI 2-sided [-6.5 to 4.3] — The mean difference is an adjusted Least Square Mean
Statistical Analysis 2: Comparison: Cohort 2; Change from baseline to week 12 in the peabody picture vocabulary test age-based standard score; Test type: Other — [test comment as in outcome 19, analysis 1]; p = 0.9546, ANCOVA; Mean Difference (Net) = -0.1, 95% CI 2-sided [-5.5 to 5.2] — The mean difference is an adjusted Least Square Mean

20. Secondary Outcome: Biomarker - Lymphocyte GSK3β Levels and Activity
Description: Total levels of GSK3β protein was determined via x-MAP technology in a Luminex 200 platform using the AKT Pathway Total Multispecies 7-Plex Panel from ThermoFisher Scientific.
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: microgram per microliter
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 8
microgram per microliter | 1.42 (0.81) | 1.95 (0.79)

ADVERSE EVENTS:
Time Frame: Consent to end of study, up to 14 weeks
Description: SAEs were collected from the time of informed consent. Non-serious AEs were collected from the time of single-blind dosing. Any non-serious medical occurrences occurring between Screening (visit 1) and Run in (visit 2) were recorded as Medical/Surgical History. Any non-serious signs and symptoms occurring between Screening (visit 1) and Run in (visit 2) were recorded and classified as baseline signs and symptoms.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 8/8 | 6/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=8)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system cyst (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Post-tussive vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Axillary mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (4)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to publish study results from his/her specific site. However, any publication that includes AMO Pharma confidential information cannot be submitted for publication without AMO Pharma's prior written approval.

DOCUMENTS (2):
  • Study Protocol (2017-01-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT02858908/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT02858908/SAP_001.pdf